CLINICAL TRIAL: NCT00717873
Title: Evaluation of High-Frequency Chest Wall Oscillation Using the Vest Airway Clearance System Compared to Conventional Chest Physical Therapy at Barnes-Jewish Hospital
Brief Title: Evaluation of High-Frequency Chest Wall Oscillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hill-Rom (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-0080
Record Dates: First submitted 2008-07-01; First posted 2008-07-18 (Estimated); Results first posted 2015-09-25 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-07

CONDITIONS: Airway Secretion Clearance
Keywords: Mucus Clearance; Secretion Clearance; HFCWO

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HFCWO Arm (Experimental): Airway clearance provided by the Vest Airway Clearance System
  Interventions: Device: Airway clearance Device
- CPT Arm (No Intervention): Airway clearance provided by manual CPT

INTERVENTIONS:
Device: Airway clearance Device — Provided by the Vest Airway clearance system
  Arms: HFCWO Arm

SUMMARY:
To compare the outcomes of patients treated with the Vest and conventional chest physiotherapy to determine if the Vest provides equivalent therapy

ELIGIBILITY:
Inclusion Criteria:

* Acute or chronic disease requiring secretion mobilization as per hospital protocol

Exclusion Criteria:

* Absolute contraindications for positional changes
* Absolute contraindications for chest percussion
* Women visibly pregnant
* Previous enrollment in study
* Previous CPT or Vest treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2008-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darnetta Clinkscale, RRT, Principal Investigator — Barnes-Jewish Hospital
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Derived] Morrison L, Milroy S. Oscillating devices for airway clearance in people with cystic fibrosis. Cochrane Database Syst Rev. 2020 Apr 30;4(4):CD006842. doi: 10.1002/14651858.CD006842.pub5. PMID 32352564
- [Derived] Clinkscale D, Spihlman K, Watts P, Rosenbluth D, Kollef MH. A randomized trial of conventional chest physical therapy versus high frequency chest wall compressions in intubated and non-intubated adults. Respir Care. 2012 Feb;57(2):221-8. doi: 10.4187/respcare.01299. Epub 2011 Jul 12. PMID 21762564

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HFCWO Arm | CPT Arm
Started | 46 | 59
Completed | 46 | 59
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HFCWO Arm | CPT Arm | Total
Number analyzed (Participants) | 46 | 59 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (18) | 45 (18) | 44 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 33 | 50
  Male | 29 | 26 | 55

OUTCOME MEASURES:

1. Primary Outcome: Hospital Length of Stay
Description: an average of 10 days
Time Frame: Admission to Discharge
Measure: Mean (Standard Deviation); unit: days
Arm/Group | HFCWO Arm | CPT Arm
Number analyzed (Participants) | 46 | 59
days | 2.95 (1.01) | 5.45 (1.84)

ADVERSE EVENTS:
Arm/Group | HFCWO Arm | CPT Arm
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/59
Other Adverse Events (participants affected / at risk) | 0/46 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No